CLINICAL TRIAL: NCT06669702
Title: EXercise As an Anti-inflammatory Treatment in Axial Spondyloarthritis (axSpA) for Patients Taking Biologic Therapy: a Proof of Concept Study (ExTASI-B).
Brief Title: EXercise Therapy in Axial SpA, Inflammation and Biologic Therapy (ExTASI-B)
Acronym: ExTASI-B
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Loughborough University (Other)
Collaborators: University Hospitals, Leicester (Other)
Responsible Party: Principal Investigator, Nicolette Bishop, Professor, Loughborough University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRAS project ID: 333667
Record Dates: First submitted 2024-10-30; First posted 2024-11-01 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Axial Spondyloarthrithis; Inflammatory Diseases; Arthritis
Keywords: Exercise; Inflammation; Immunosenescence
MeSH Terms: conditions — Arthritis; Motor Activity; Inflammation

STUDY DESIGN:
Intervention Model Description: Random allocation into either a control group or an exercise group (12-weeks of home based exercise).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (No Intervention): Healthy controls
- Exercise (Experimental): 12-weeks of home based exercise involving 30 minutes of brisk walking on 5 days per week.
  Interventions: Behavioral: 12-week home based exercise
- Routine care (Experimental): Routine care
  Interventions: Behavioral: Routine care

INTERVENTIONS:
Behavioral: 12-week home based exercise — Patients allocated to the exercise arm will be prescribed a home-based walking exercise programme consisting of 30 minutes of walking on 5 days per week at an rating of perceived exertion in the range of 12-14 (somewhat hard). Each patient's heart rate range will be established during the baseline exercise test by recording the heart rate response at the required RPE target range. This will be provided to each patient to use in conjunction with the activity monitor they will be given to wear on their non-dominant wrist. The monitor reports heart rate and records daily steps, distance and activity duration.
  Participants can break down the exercise time in a way that suits their time, i.e., they can do 3 × 10 minutes, 2 × 15 minutes, etc.
  Arms: Exercise
Behavioral: Routine care — Participants in this group will continue with their current routine care and will be given a diary of exercises that they can do, which are usually given to them as part of their health care routine by physiotherapists or consultants. The diary has information about yoga-like stretching practices.
  Arms: Routine care

SUMMARY:
The goal of this randomised controlled trial study is to investigate whether exercise (brisk walking, equal to 13 on a rating of perceived exertion scale; somewhat hard) can be used as an adjuvant therapy for people living with axial spondyloarthritis and taking biologic medications to further improve their quality of life and lower their symptoms and disease burden. The main questions it aims to answer are:

Does a 12-week structured home-based aerobic exercise intervention have a favourable effect on markers of immune-mediated inflammation and symptom severity?

As a secondary aim and outcome, this study will investigate:

* The acceptability of this intervention using questionnaires with free text boxes and one-to-one semi-structured interviews in a subset (50%) of participants (Q-ExTASI-B substudy).
* The effect of the home-based intervention on circulating markers of cardiometabolic health, anthropometrical measures, and immune markers that associate with systemic inflammation.
* The effect of the home-based intervention on objective measures of physical function and exercise tolerance

The study will compare the data of a healthy group with that of people living with axial spondyloarthritis. Within the patient population, 20 of the individuals will be allocated to the exercise group (randomly), and 20 will be allocated to the usual care group. In the exercise group, participants will be asked to do 30 minutes of brisk walking five days a week for 12 weeks, and they will be visiting Loughborough University every four weeks to provide blood samples and fill out questionnaires. Participants in the usual care group will continue with their current care routine and will visit the study site to provide blood samples and questionnaire data every 4 weeks. The data from all axSpA patients will be compared to healthy controls, and subgroup analysis will be conducted to investigate the difference between the exercise group and the usual care group.

DETAILED DESCRIPTION:
Over 200,000 people in the UK have axial spondyloarthritis. In 80% of cases the condition begins in the second or third decade of life. Exercise is encouraged as an essential treatment of axial spondyloarthritis (axSpA), with the potential to both promote well-being, increase flexibility and range of movement, improve posture and reduce stiffness and pain. axSpA is an inflammatory arthritis and raised levels of indicators ('markers') of this inflammatory process (e.g. CRP) can be detected in the blood of patients. These markers are released as a consequence of the condition, but some, such as TNF-alpha and interleukin-17 (IL-17), also promote further disease development. In other inflamed patient groups we have shown that regular exercise (brisk walking) can lower the levels of these pro-inflammatory markers in the blood and increase levels of anti-inflammatory markers, independently of weight loss. Despite axSpA being an inflammatory condition with prescribed medication focused on reducing inflammation there are no studies that have assessed the potential of exercise to act as an anti-inflammatory adjuvant to biologic therapy in axSpA. This research will investigate the effect of 12 weeks of a home-based walking exercise intervention on measures of systemic inflammation and body composition, well-being and measures of disease activity using established and validated methods in 20 axSpA patients on regular biologic therapy and compare this group with 20 patients on regular biologic therapy who carry on with their standard care and normal levels of activity. Also, a baseline comparison will be conducted between a group of 20 healthy individuals and axSpA patients (40).This proof-of-concept study will determine the potential of exercise as an adjuvant anti-inflammatory treatment for patients with axSpA taking biologic medication.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of axSpA by a consultant rheumatologist
* Age=/>18 years old
* Without other significant cardiovascular comorbidities
* Receiving stable dose biologic treatment
* Able to commit to the time demands of the study

Exclusion Criteria:

* Unable to undertake exercise due to physical or psychological barriers
* Presence of hip or peripheral joint disease
* Contraindication to exercise training (American College of Sports Medicine guidelines)
* Excessively active (score of high on IPAQ)
* Unable to communicate sufficiently in English
* Female participants who are pregnant, lactating, or planning pregnancy during the course of the study.
* Inability to give informed consent or comply with testing and training protocol for any reason.
* Presence of chronic anaemia (haemoglobin less than 13.5 g/dL for men; less than 12.0 g/dL for women; or haematocrit less than 41.0% in men, less than 36.0% in women.
* Co-morbidity that the research team determine to be a contraindication to involvement

Inclusion and exclusion criteria of healthy controls:

Inclusion Criteria:

* Aged between 18 years old and 65 years old
* Not taking any long-term medication that affects inflammation or immune-mediated inflammation.
* Free from infection or infection symptoms

Exclusion criteria:

The participant may not enter the study if ANY of the following apply:

* Unable to undertake exercise due to physical or psychological barriers
* Excessively active (score of high on IPAQ)
* Unable to communicate sufficiently in English
* Female participants who are pregnant, lactating, or planning pregnancy during the course of the study.
* Inability to give informed consent or comply with testing and training protocol for any reason.
* Have been diagnosed with or are aware of at least one of the following health issues:
* Immune system disorder
* Cardiovascular and/or cardiometabolic diseases, including but not limited to high blood pressure, high triglycerides and/or cholesterol levels, diabetes mellitus, etc.
* Any chronic health condition that affects one's ability to partake in physical activity
* Musculoskeletal injury that affects one's ability to partake in physical activity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Changes in spinal pain before (week 0 - baseline), and during (weeks 4, 8, and 12), the 12-week home based exercise intervention. | 0, 4, 8, 12 weeks
  Using the validated visual analogue scale for spinal pain. The scale consists of a straight line with the end points defining extreme limits 'no spinal pain' and 'spinal pain as bad as it could be'. The line is 10cm in length (0cm point representing no pain, 10cm point representing pain as bad as it could be). A score of 0-10 is given depending on where the patient marks the line (5cm representing a score of 5). The higher the score, the worse the spinal pain.
Changes in inflammatory monocyte phenotypes before (week 0 - baseline), and during (weeks 4, 8, and 12), the 12-week home based exercise intervention | 0, 4, 8, 12, weeks.
  Expression of receptors associated with inflammatory activity and stimulated cell inflammatory cytokine release. This will be analysed via flow cytometry.
Changes in ankylosing spondylitis disease activity before (week 0 - baseline), and during (weeks 4, 8, and 12), the 12-week home based exercise intervention. | 0, 4, 8, 12, weeks.
  Using the validated Bath Ankylosing Spondylitis Disease Activity Index (BASDAI). The BASDAI consists of a 0-10 score (0 being no problem and 10 being the worst problem) which is used to answer 6 questions on fatigue, spinal pain, joint pain, tenderness, morning stiffness duration, and morning stiffness severity. To give each symptom equal weighting, the mean (average) of the two scores relating to stiffness is taken. The resulting 0 to 50 score is divided by 5 to give a final 0 - 10 BASDAI score. The higher the score, the higher the activity of disease.
Changes in characteristics of T-cell cell phenotypes (senescence) before (week 0 - baseline), and during (weeks 4, 8, and 12), the 12-week home based exercise intervention | 0, 4, 8, 12, weeks.
  Expression of receptors associated with senescence. This will be analysed via flow cytometry

SECONDARY OUTCOMES:
Changes in tumor necrosis factor-alpha blood concentrations before (week 0 - baseline), and during (weeks 4, 8, and 12), the 12-week home based exercise intervention. | 0, 4, 8, 12, weeks
Changes in interleukin-6 blood concentrations before (week 0 - baseline), and during (weeks 4, 8, and 12), the 12-week home based exercise intervention. | 0, 4, 8, 12, weeks
Changes in stimulated cytokine concentration released from isolated Peripheral blood mononuclear cells (PBMCs) before (week 0 - baseline), and after (weeks 12), the 12-week home based exercise intervention. | 0,12, weeks
  PBMCs will be isolated using centrifuge and then cultured with PMA ionomycin to stimulate cytokine release. Concentrations of released inflammatory cytokines will be compared to a control culture (no PMA ionomycin stimulation).
Changes in the symptom burden of ankylosing spondylitis before (week 0 - baseline), and during (weeks 4, 8, and 12), the 12-week home based exercise intervention. | 0, 4, 8, 12, weeks.
  Using the validated Bath Ankylosing Spondylitis Functional Index (BASFI). The index assesses the functional limitation in patients with ankylosing spondylitis by asking the patient about symptom burden. The index consists of 10 questions evaluating how hard the patient finds situations i.e 'how difficult is it to put on your socks?' A score of 0 represents easy, and a score of 10 represents impossible. The mean (average) of the 10 questions is used to assign a symptom burden score of 0-10. The higher the score, the higher the symptom burden caused by ankylosing spondylitis.
Changes in work productivity before (week 0 - baseline), and during (weeks 4, 8, and 12), the 12-week home based exercise intervention. | 0, 4, 8, 12, weeks.
  Using the validated work productivity and activity impairment questionnaire (WPAI:GH). The questionnaire asks about the effect of health problems on the ability to work and perform regular activities. The questionnaire outcome is expressed as an impairment percentage, with higher numbers indicating greater impairment and less productivity.
Changes in subjective physical activity before (week 0 - baseline), and after (week 12) the 12-week home based exercise intervention. | 0, 12, weeks.
  Measured from the international physical activity questionnaire (IPAQ). The IPAQ asks 27 questions on physical activity (PA).
  Those who score 'high' engage in: 1) vigorous activity on at least 3 days achieving a total PA of at least 1500 metabolic equivalent of task (MET) minutes a week - OR - 2) 7 or more days of any combination of walking, moderate intensity or vigorous intensity activities achieving a minimum total PA of at least 3000 MET minutes per week.
  Those who score 'moderate' engage in: 1) 3 or more days of vigorous intensity activity and/or walking of at least 30 minutes per day - OR - 2) 5 or more days of moderate intensity activity and/or walking of at least 30 minutes per day
  - OR - 3) 5 or more days of any combination of walking, moderate intensity, or vigorous intensity activities achieving a minimum total PA of at least 600 MET minutes per week.
  Those who score 'low' do not fit the criteria of either the moderate or high levels of PA.
Adherence to biologic medicines before (week 0 - baseline), and during (week 4, 8, 12) the 12-week home based exercise intervention. | 0, 4, 8, 12 weeks.
  Using the validated Compliance Questionnaire Rheumatology (CQR). The CQR measures adherence to prescribed exercise or medication regimens in patients with rheumatic diseases, including ankylosing spondylitis. It consists of 19 items scored on a Likert scale, where 1 indicates "strongly disagree" and 4 indicates "strongly agree." The responses are combined to calculate a compliance score ranging from 0-100, with higher scores indicating better adherence to the intervention.
Changes in quality of life of the patients before (week 0 - baseline), and during (weeks 4, 8, 12) the 12-week home based exercise intervention. | 0, 4, 8, 12 weeks.
  Using the validated Ankylosing Spondylitis Quality of Life (ASQoL) questionnaire. The ASQoL is a disease-specific instrument designed to measure the impact of ankylosing spondylitis on a patient's quality of life. It consists of 18 yes/no questions, with each "yes" response contributing to a total score. Scores range from 0 to 18, with higher scores indicating a greater impact of the disease on the patient's quality of life.
Changes in the general health-related quality of life before (week 0 - baseline), and during (weeks 4, 8, and 12), the 12-week home-based exercise intervention. | 0, 4, 8, 12 weeks.
  Using the EuroQol 5-Dimension (EQ-5D) questionnaire. The EQ-5D is a standardized instrument used to measure health-related quality of life across five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is scored on a scale of 1 to 5, representing different levels of severity, with a total score reflecting the overall health status. Additionally, a visual analogue scale (VAS) is used to rate the patient's perceived health on a scale from 0 to 100, with higher scores indicating better health-related quality of life.
Changes in overall health status before (week 0 - baseline), and during (weeks 4, 8, and 12), the 12-week home-based exercise intervention. | 0, 4, 8, 12 weeks.
  Using the Medical Outcomes Study 36-Item Short Form Health Survey (SF-36). The SF-36 assesses overall health status across eight domains: physical functioning, role limitations due to physical health, bodily pain, general health perceptions, vitality (energy/fatigue), social functioning, role limitations due to emotional problems, and mental health. Each domain is scored on a scale from 0 to 100, with higher scores indicating better health and less limitation in that area. The SF-36 provides a comprehensive view of both physical and mental health.
Changes in daytime sleepiness before (week 0 - baseline), and during (weeks 4, 8, and 12), the 12-week home-based exercise intervention. | 0, 4, 8, 12 weeks.
  Using the Epworth Sleepiness Scale (ESS). The ESS is a validated questionnaire that assesses daytime sleepiness by asking patients to rate their likelihood of falling asleep in eight common situations, such as sitting and reading or watching television. Each situation is rated on a scale from 0 (would never doze) to 3 (high chance of dozing), with a total score ranging from 0 to 24. Higher scores indicate greater levels of daytime sleepiness, which may affect daily functioning.
Changes in night time sleep quality before (week 0 - baseline), and during (weeks 4, 8, and 12), the 12-week home-based exercise intervention. | 0, 4, 8, 12 weeks.
  Using the Pittsburgh Sleep Quality Index (PSQI). The PSQI measures sleep quality and disturbances over a 1-month period. It consists of 19 items grouped into seven components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. Each component is scored from 0 to 3, and the component scores are summed to produce a global score ranging from 0 to 21. Higher scores indicate poorer sleep quality.
Changes in gastrointestinal symptoms before (week 0 - baseline), and during (weeks 4, 8, and 12), the 12-week home-based exercise intervention. | 0, 4, 8, 12 weeks.
  Using the Crohn's and Ulcerative Colitis Questionnaire-8 (CUCQ-8). The CUCQ-8 is a short, validated questionnaire used to assess the symptom burden in patients with Crohn's disease and ulcerative colitis. It consists of eight items that evaluate key symptoms such as abdominal pain, bowel urgency, and the frequency of bowel movements. Each item is scored on a scale from 0 (no symptoms) to 4 (severe symptoms), with a total score ranging from 0 to 32. Higher scores indicate a greater burden of gastrointestinal symptoms.
Changes in physical function before (week 0 - baseline), and after (week 12) the 12-week home based exercise intervention. | 0, 12 weeks.
  Sit to stand-5 test (STS-5). The test consists of going from a seated to a standing position 5 times as quickly as possible.
Changes in secondary physical function before (week 0 - baseline), and after (week 12) the 12- week home based exercise intervention. | 0, 12 weeks.
  Sit to stand-60 test (STS-60). The test consists of going from a seated to a standing position as many times as possible within 60 seconds.
Changes in exercise capacity before (week 0 - baseline), and after (week 12), the 12-week home-based exercise intervention. | 0, 12 weeks.
  Using the Incremental Shuttle Walk Test (ISWT). The ISWT is a standardised field test used to assess functional exercise capacity. Patients walk back and forth along a 10-meter course, with the walking speed progressively increasing according to audio signals. The test continues until the patient is unable to keep up with the pace, becomes breathless, or reaches 85% of their age-relative maximum heart rate. The total distance walked is recorded and used to evaluate changes in exercise capacity. Greater distances indicate improved functional capacity and physical fitness.
Changes in body mass before (week 0 - baseline), and during (weeks 4, 8, and 12) the 12-week home based exercise intervention. | 0, 4, 8, 12 weeks.
  Kilograms
Changes in height before (week 0 - baseline), and during (weeks 4, 8, and 12) the 12-week home based exercise intervention. | 0, 4, 8, 12 weeks.
  Centimetres
Changes in waist circumference before (week 0 - baseline), and during (weeks 4, 8, and 12) the 12-week home based exercise intervention. | 0, 4, 8, 12 weeks.
  Centimetres
Changes in hip circumference before (week 0 - baseline), and during (weeks 4, 8, and 12) the 12-week home based exercise intervention. | 0, 4, 8, 12 weeks.
  Centimetres
Changes in body fat percentage before (week 0 - baseline), and during (weeks 4, 8, and 12) the 12-week home based exercise intervention. | 0, 4, 8, 12 weeks.
  Via tanita body composition scales (bio electrical impedance analysis).
Sedentary activity minutes per day | 7 days in the 2 week period prior to baseline assessment.
  All participants will wear an Actigraph activity monitor on their non-dominant wrist to record physical activity for 7 days in the two weeks before the baseline assessment visit to characterise physical activity levels.
  The Freedson (1998) activity monitor counts per minute cut points will be used to quantify minutes per day spent sedentary.
Light physical activity minutes per day | 7 days in the 2 week period prior to baseline assessment.
  All participants will wear an Actigraph activity monitor on their non-dominant wrist to record physical activity for 7 days in the two weeks before the baseline assessment visit to characterise physical activity levels.
  The Freedson (1998) activity monitor counts per minute cut points will be used to quantify minutes per day spent in light activity.
Moderate to vigorous physical activity minutes per day | 7 days in the 2 week period prior to baseline assessment.
  All participants will wear an Actigraph activity monitor on their non-dominant wrist to record physical activity for 7 days in the two weeks before the baseline assessment visit to characterise physical activity levels.
  The Freedson (1998) activity monitor counts per minute cut points will be used to quantify minutes per day spent in moderate to vigorous physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Arumugam Moorthy, Dr, Principal Investigator — University Hospitals, Leicester
Locations (2):
- United Kingdom (2):
  - Loughborough University, National Centre for Sport and Exercise Medicine, Loughborough, Leicestershire
  - University Hospitals of Leicester NHS trust, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
According to informed consent, no IPD will be shared with any external parties.

REFERENCES:
- [Background] Roberts MJ, Hamrouni M, Linsley V, Moorthy A, Bishop NC. Exercise as an anti-inflammatory Therapy in Axial Spondyloarthritis Therapeutic Intervention (EXTASI) study: a randomized controlled trial. Rheumatol Adv Pract. 2024 May 11;8(2):rkae062. doi: 10.1093/rap/rkae062. eCollection 2024. PMID 38854418
- [Background] Dungey M, Young HML, Churchward DR, Burton JO, Smith AC, Bishop NC. Regular exercise during haemodialysis promotes an anti-inflammatory leucocyte profile. Clin Kidney J. 2017 Dec;10(6):813-821. doi: 10.1093/ckj/sfx015. Epub 2017 Mar 27. PMID 29225811
- [Background] Minuzzi LG, Rama L, Bishop NC, Rosado F, Martinho A, Paiva A, Teixeira AM. Lifelong training improves anti-inflammatory environment and maintains the number of regulatory T cells in masters athletes. Eur J Appl Physiol. 2017 Jun;117(6):1131-1140. doi: 10.1007/s00421-017-3600-6. Epub 2017 Apr 8. PMID 28391394
- [Background] Viana JL, Kosmadakis GC, Watson EL, Bevington A, Feehally J, Bishop NC, Smith AC. Evidence for anti-inflammatory effects of exercise in CKD. J Am Soc Nephrol. 2014 Sep;25(9):2121-30. doi: 10.1681/ASN.2013070702. Epub 2014 Apr 3. PMID 24700875
- [Background] Gleeson M, Bishop NC, Stensel DJ, Lindley MR, Mastana SS, Nimmo MA. The anti-inflammatory effects of exercise: mechanisms and implications for the prevention and treatment of disease. Nat Rev Immunol. 2011 Aug 5;11(9):607-15. doi: 10.1038/nri3041. PMID 21818123
- [Background] Pecourneau V, Degboe Y, Barnetche T, Cantagrel A, Constantin A, Ruyssen-Witrand A. Effectiveness of Exercise Programs in Ankylosing Spondylitis: A Meta-Analysis of Randomized Controlled Trials. Arch Phys Med Rehabil. 2018 Feb;99(2):383-389.e1. doi: 10.1016/j.apmr.2017.07.015. Epub 2017 Aug 30. PMID 28860095
- [Background] Beavers KM, Brinkley TE, Nicklas BJ. Effect of exercise training on chronic inflammation. Clin Chim Acta. 2010 Jun 3;411(11-12):785-93. doi: 10.1016/j.cca.2010.02.069. Epub 2010 Feb 25. PMID 20188719
- [Background] Borg G, Hassmen P, Lagerstrom M. Perceived exertion related to heart rate and blood lactate during arm and leg exercise. Eur J Appl Physiol Occup Physiol. 1987;56(6):679-85. doi: 10.1007/BF00424810. PMID 3678222
- [Background] Highton PJ, White AEM, Nixon DGD, Wilkinson TJ, Neale J, Martin N, Bishop NC, Smith AC. Influence of acute moderate- to high-intensity aerobic exercise on markers of immune function and microparticles in renal transplant recipients. Am J Physiol Renal Physiol. 2020 Jan 1;318(1):F76-F85. doi: 10.1152/ajprenal.00332.2019. Epub 2019 Nov 18. PMID 31736354
- [Background] Billany RE, Smith AC, Stevinson C, Clarke AL, Graham-Brown MPM, Bishop NC. Perceived barriers and facilitators to exercise in kidney transplant recipients: A qualitative study. Health Expect. 2022 Apr;25(2):764-774. doi: 10.1111/hex.13423. Epub 2022 Jan 10. PMID 35014114
- [Background] Schafer JL. Multiple imputation: a primer. Stat Methods Med Res. 1999 Mar;8(1):3-15. doi: 10.1177/096228029900800102. PMID 10347857